CLINICAL TRIAL: NCT01631253
Title: The Impact on Ovarian Reserve After Single-port, Two-port, or Four-port Access Laparoscopic Ovarian Cyst Enucleation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Seok Ju Seong, Principal Investigator, CHA University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPA001
Record Dates: First submitted 2012-06-26; First posted 2012-06-29 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Ovarian Cyst
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- single-port access laparoscopic ovarian cyst enucleation (Active Comparator): Procedure: Operative laparoscopic ovarian cyst enucleation was performed only through an umbilical single port. ( 2 cm longitudinal incision was made within the umbilicus and an wound retractor (Alexis Wound Retractor XS) was inserted into the wound opening. A surgical glove with three 5mm trocars inserted into three fingers was draped around the rim of the wound retractor.)
  Interventions: Procedure: Laparoscopic ovarian cyst enucleation
- two-port laparoscopic access ovarian cyst enucleation (Active Comparator): Procedure: Operative access laparoscopic ovarian cyst enucleation was performed using an umbilical single port ( 2 cm longitudinal incision was made within the umbilicus and an wound retractor (Alexis Wound Retractor XS) was inserted into the wound opening. A surgical glove with two 5mm trocars inserted into two fingers was draped around the rim of the wound retractor.) and one 5-mm trocar in the lower abdomen.
  Interventions: Procedure: Laparoscopic ovarian cyst enucleation
- four-port access laparoscopic ovarian cyst enucleation (Active Comparator): Procedure: : Operative laparoscopic ovarian cyst enucleation was performed through insertion of a 12-mm subumbilical trocar and three 5-mm trocars in the lower abdomen.
  Interventions: Procedure: Laparoscopic ovarian cyst enucleation

INTERVENTIONS:
Procedure: Laparoscopic ovarian cyst enucleation

SUMMARY:
The purpose of this study is to investigate the impact on ovarian reserve after single- port, two-port, or four-port access laparoscopic ovarian cyst enucleation based on serum anti mullerian hormone change.

DETAILED DESCRIPTION:
With the recent development of surgical instruments techniques, minimally invasive surgery is more feasible in various field of surgery. Laparoscopic surgery has potential benefit of decreased patient discomfort, short hospital stay, superior cosmetic results and decreased convalescence time. Recently, various efforts have been continued for minimally invasive surgery, one of the recently emerging concepts is single port surgery. Several studies have demonstrated that single-port laparoscopic surgery is feasible and safe in gynecology.

However, some limits could be occurred, such as the occurrence of less freedom degrees between the instruments and limits surgical vision, thus limiting surgeon's movements. So, two-port laparoscopy combined access through umbilical and additional suprapubic incision have been used and reported. In case of single port access laparoscopic ovarian cyst enucleation, due to limits of surgeon's movements, cyst enucleation or bipolar electrocoagulation of the ovarian parenchyma adversely affected ovarian function.

Some studies reported that after laparoscopic cyst enucleation, there had been shown marked reduction of ovarian function compared with surgery by laparotomy. Therefore we attempt to investigate the impact of single port laparoscopy that have limits of surgical procedures on ovarian reserve after ovarian cyst enucleation.

To evaluate ovarian reserve change, we will use the anti-mullerian hormone. It is produced by granulosa cells of preantral and small antral follicles and has been recently acknowledged as the useful, reliable, and sensitive hormonal serum marker of the ovarian primordial follicle pool. In addition, the AMH level represents a stronger independent marker of ovarian reserve without significant fluctuation during the menstrual cycle, which progressively decreases with age.

Therefore, this prospective study is performed to compare the differences in ovarian reserve after single-port, two-port, or four-port access laparoscopic ovarian cyst enucleation based on serum anti mullerian hormone change. Serum anti mullerian hormone is measured at preoperative and at postoperative 1week, 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-45 years Ultrasound
* CT, MRI diagnosis as ovarian cyst , need to cyst enucleation
* Size of cyst : between 3cm and 10cm
* Regular menstrual cycles defined as cycle length between 25 and 35 days
* Agreement to be enrolled in the study.

Exclusion Criteria:

* Previous ovarian surgery
* suspicious of malignancy
* Postmenopause
* Use of oral contraceptive drug, GnRH agonist /antagonist, or other drugs related with ovarian function in last 3 months
* Known endocrine disorder

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Preoperative and postoperative changes in anti-mullerian hormone level | preoperative, postoperative at 1week, 1 and 3 months
  The primary outcome of our study is the impact on ovarian reserve determined by AMH after the application of the three laparoscopic techniques for the treatment of ovarian cyst.In all study patients, at preoperation and 1 week, 1 month, 3 month after operation, AMH is serially measured.

SECONDARY OUTCOMES:
postoperative pain scores

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam CHA medical center, Seoul, Gamnamgu, South Korea

REFERENCES:
- [Derived] Yoon BS, Kim YS, Seong SJ, Song T, Kim ML, Kim MK, Paek JY. Impact on ovarian reserve after laparoscopic ovarian cystectomy with reduced port number: a randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2014 May;176:34-8. doi: 10.1016/j.ejogrb.2014.02.025. Epub 2014 Feb 20. PMID 24630293